CLINICAL TRIAL: NCT00751452
Title: Evaluation of Citrullinemia as a Marker of Bowel Damage After Allogeneic Bone Marrow Transplantation in Children
Brief Title: Citrulline Allo. Evaluation of Citrullinemia as a Marker of Bowel Damage After Allogeneic Bone Marrow Transplantation in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Merlin Etienne, CHU Clermont-Ferrand
Other Study IDs: CHU-0040
Record Dates: First submitted 2008-09-09; First posted 2008-09-12 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Benign Disease
Keywords: Children; Allogeneic bone marrow transplantation; Intestinal damage; Citrulline; Graft versus Host Disease; 0 to 18 years old
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
determine the interest of the dosage of citrullinemia to monitor the bowel damage after allogeneic bone marrow transplantation in children.

DETAILED DESCRIPTION:
30 children included. Dosage of citrullinemia on day -7, day 0 and every week up to 100 days after BMT. Histological examination and extensive infectious screening in case of persistent digestive symptoms (more than 3 days).

Two groups of patients regarding on digestive involvement. Comparison of the values of citrullinemia between these two groups.

ELIGIBILITY:
Inclusion Criteria:

* 0 to 18 years
* allogeneic bone marrow transplantation for malignant or benign disease
* affiliation to French sécurité sociale
* parent's consent

Exclusion Criteria:

* severe gastro-intestinal involvement before transplant
* previous digestive surgery

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: screening
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Citrullinemia (weekly) | weekly

SECONDARY OUTCOMES:
Gastro-intestinal complications in children following allogeneic bone marrow transplantation | following allogenic bone marrow transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Merlin Etienne, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Etienne MERLIN, Clermont-Ferrand, France